CLINICAL TRIAL: NCT03429296
Title: Prospective, Randomized Study Aiming to Assess the Benefit of Autohypnosis Learning in the Care of Patients Treated by Adjuvant Chemotherapy for Colorectal or Breast Cancer.
Brief Title: Autohypnosis and Cancerology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Collaborators: TIMC-IMAG (Other); AG2R La Mondiale (Other); GEFLUC (Unknown); Espoir Isère Cancer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/12-SBO-GHMG
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer; Breast Cancer
Keywords: Cancer; Autohypnosis; Quality of life
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Zelen : patients will be randomized according to the Zelen randomization design (as described in "Zelen M. Randomized consent designs for clinical trials: An update. Stats in Med. 1990;9:645-656")
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autohypnosis learning (Experimental): In this arm, patients are taught autohypnosis during sessions in groups of 3 to 6 with a qualified hypnotherapist. Sessions are set every two weeks, for a total of 6 sessions. Individual sessions are possible for patients who missed a session.
  Interventions: Other: Autohypnosis learning
- Standard of care (No Intervention): In this arm, patients are not taught autohypnosis and are treated according to standard of care.

INTERVENTIONS:
Other: Autohypnosis learning — Patients are taught how to do auto-hypnosis by an hypnotherapist before all along their chemotherapy.
  Arms: Autohypnosis learning

SUMMARY:
Therapeutical hypnosis is proven to be an effective medical support to chemotherapy: it was shown that it can reduce the pain, anxiety, fatigue felt by the patient.

Yet, hypnosis requires the presence of an hypnotherapist, which is why auto-hypnosis could be an efficient alternative to handle the side effects of chemotherapy.

In this study, colorectal cancer and breast cancer patients are either taught auto-hypnosis or are taken in standard care for their chemotherapy.

The life quality score (QLQC30) assessed during and after chemotherapies will determine if auto-hypnosis is a good medical support in chemotherapies' adverse effects management.

The proven benefices of auto-hypnosis in the handling of the side effects of chemotherapies could improve the quality of life of cancer affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Age superior or equal to 18 years old
* Colorectal or breast cancer history, treated by surgery and that should undergo an adjuvant chemotherapy

  * In the case of breast cancer, adjuvant chemotherapy must involve anthracyclines
* ECOG performance score < 3
* Patient must be affiliated or beneficiary of social security or any similar regime

Exclusion Criteria:

* Patients already included in another interventional clinical research protocol
* Patients unable to proceed to hypnosis treatment due to their speech limitations (poor comprehension and expression of french, deafness, mental illness)
* Patients protected by French law from clinical inclusion ( pregnant, in labour, breastfeeding, legally protected, under judiciary or administrative liberty deprivation...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
>20% increase of the EORTC QLQC30 score (annexe 1) at the third week after the last chemotherapy session in the auto-hypnosis arm compared to the standard care arm. | 3 weeks after the last chemotherapy session
  At the third week after the last chemotherapy session, patients answer the quality of life survey (EORTC QLQC30). Arms' mean score are compared, a minimal difference of 21% is needed for statistical significance.

SECONDARY OUTCOMES:
Evaluation of auto-hypnosis effects on the life quality and global health of patients at short, mid, and long term. | 3rd week and 6 month after the last treatment and either one in two chemotherapy sessions, or each chemotherapy session if XELOX treatment
  Patients answer the quality of life survey (EORTC QLQC30) one in two chemotherapy session, or each session for XELOX therapy.
Evaluation of auto-hypnosis effects on different components of quality of life. | 3rd week and 6 month after the last treatment and either one in two chemotherapy sessions, or each chemotherapy session if XELOX treatment
  Quantitative evaluation of QLQ-C30 subdomains
Evaluation of auto-hypnosis effects on different components of quality of life specific to breast cancer | 3rd week and 6 month after the last treatment and either one in two chemotherapy sessions, or each chemotherapy session if XELOX treatment
  Quantitative evaluation of QLQ-BR23 scores
Evaluation of auto-hypnosis effects on different components of quality of life specific to colorectal cancer. | 3rd week and 6 month after the last treatment and either one in two chemotherapy sessions, or each chemotherapy session if XELOX treatment
  Quantitative evaluation of QLQ-CR29 scores
Evaluation of auto-hypnosis effects on drug consumption. | 3rd week and 6 month after the last treatment and either one in two chemotherapy sessions, or each chemotherapy session if XELOX treatment
  Patients answer a survey about their consumption of different type of drugs : pain-killers, antiemetics, anxiolytics, sleeping drugs.
Evaluation of auto-hypnosis effects on fatigue. | 3rd week and 6 month after the last treatment and either one in two chemotherapy sessions, or each chemotherapy session if XELOX treatment
  Evaluation of fatigue score MFI-20
Evaluation of auto-hypnosis impact on anxiety and/or depression. | 3rd week and 6 month after the last treatment and either one in two chemotherapy sessions, or each chemotherapy session if XELOX treatment
  Evaluation of HADS score
Evaluation of auto-hypnosis impact on the global medical handling of their cancer. | 3rd week and 6 month after the last treatment
  Numerical scale of satisfaction survey (from 0 to 10) 0 will mean "very unsatisfied" and 10 will mean "very satisfied".
Evaluation of patient's satisfaction about auto-hypnosis therapies. | 3rd week and 6 month after the last treatment
  Satisfaction survey about their satisfaction about auto-hypnosis therapies

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe hospitalier Mutualiste de Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faivre J, Grosclaude P, Launoy G, Arveux P, Raverdy N, Menegoz F, Pienkowski P, Schaffer P, Daures JP, De Vathaire F. [Digestive cancers in France. Geographic distribution and estimation of national incidence]. Gastroenterol Clin Biol. 1997;21(3):174-80. French. PMID 9161491
- [Background] Edge SB, Compton CC. The American Joint Committee on Cancer: the 7th edition of the AJCC cancer staging manual and the future of TNM. Ann Surg Oncol. 2010 Jun;17(6):1471-4. doi: 10.1245/s10434-010-0985-4. PMID 20180029
- [Background] Gunderson LL, Jessup JM, Sargent DJ, Greene FL, Stewart AK. Revised TN categorization for colon cancer based on national survival outcomes data. J Clin Oncol. 2010 Jan 10;28(2):264-71. doi: 10.1200/JCO.2009.24.0952. Epub 2009 Nov 30. PMID 19949014
- [Background] Sargent DJ, Marsoni S, Monges G, Thibodeau SN, Labianca R, Hamilton SR, French AJ, Kabat B, Foster NR, Torri V, Ribic C, Grothey A, Moore M, Zaniboni A, Seitz JF, Sinicrope F, Gallinger S. Defective mismatch repair as a predictive marker for lack of efficacy of fluorouracil-based adjuvant therapy in colon cancer. J Clin Oncol. 2010 Jul 10;28(20):3219-26. doi: 10.1200/JCO.2009.27.1825. Epub 2010 May 24. PMID 20498393
- [Background] Moertel CG, Fleming TR, Macdonald JS, Haller DG, Laurie JA, Goodman PJ, Ungerleider JS, Emerson WA, Tormey DC, Glick JH, et al. Levamisole and fluorouracil for adjuvant therapy of resected colon carcinoma. N Engl J Med. 1990 Feb 8;322(6):352-8. doi: 10.1056/NEJM199002083220602. PMID 2300087
- [Background] Zaniboni A, Labianca R, Marsoni S, Torri V, Mosconi P, Grilli R, Apolone G, Cifani S, Tinazzi A. GIVIO-SITAC 01: A randomized trial of adjuvant 5-fluorouracil and folinic acid administered to patients with colon carcinoma--long term results and evaluation of the indicators of health-related quality of life. Gruppo Italiano Valutazione Interventi in Oncologia. Studio Italiano Terapia Adiuvante Colon. Cancer. 1998 Jun 1;82(11):2135-44. doi: 10.1002/(sici)1097-0142(19980601)82:113.0.co;2-u. PMID 9610692
- [Background] Efficacy of adjuvant fluorouracil and folinic acid in colon cancer. International Multicentre Pooled Analysis of Colon Cancer Trials (IMPACT) investigators. Lancet. 1995 Apr 15;345(8955):939-44. PMID 7715291
- [Background] Haller DG, Tabernero J, Maroun J, de Braud F, Price T, Van Cutsem E, Hill M, Gilberg F, Rittweger K, Schmoll HJ. Capecitabine plus oxaliplatin compared with fluorouracil and folinic acid as adjuvant therapy for stage III colon cancer. J Clin Oncol. 2011 Apr 10;29(11):1465-71. doi: 10.1200/JCO.2010.33.6297. Epub 2011 Mar 7. PMID 21383294
- [Background] Schmoll HJ, Tabernero J, Maroun J, de Braud F, Price T, Van Cutsem E, Hill M, Hoersch S, Rittweger K, Haller DG. Capecitabine Plus Oxaliplatin Compared With Fluorouracil/Folinic Acid As Adjuvant Therapy for Stage III Colon Cancer: Final Results of the NO16968 Randomized Controlled Phase III Trial. J Clin Oncol. 2015 Nov 10;33(32):3733-40. doi: 10.1200/JCO.2015.60.9107. Epub 2015 Aug 31. PMID 26324362
- [Background] Andre T, Boni C, Navarro M, Tabernero J, Hickish T, Topham C, Bonetti A, Clingan P, Bridgewater J, Rivera F, de Gramont A. Improved overall survival with oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment in stage II or III colon cancer in the MOSAIC trial. J Clin Oncol. 2009 Jul 1;27(19):3109-16. doi: 10.1200/JCO.2008.20.6771. Epub 2009 May 18. PMID 19451431
- [Background] Schmoll HJ, Twelves C, Sun W, O'Connell MJ, Cartwright T, McKenna E, Saif M, Lee S, Yothers G, Haller D. Effect of adjuvant capecitabine or fluorouracil, with or without oxaliplatin, on survival outcomes in stage III colon cancer and the effect of oxaliplatin on post-relapse survival: a pooled analysis of individual patient data from four randomised controlled trials. Lancet Oncol. 2014 Dec;15(13):1481-1492. doi: 10.1016/S1470-2045(14)70486-3. Epub 2014 Nov 12. PMID 25456367
- [Background] Association of Breast Surgery at Baso 2009. Surgical guidelines for the management of breast cancer. Eur J Surg Oncol. 2009;35 Suppl 1:1-22. doi: 10.1016/j.ejso.2009.01.008. Epub 2009 Mar 18. No abstract available. PMID 19299100
- [Background] Hammond ME. ASCO-CAP guidelines for breast predictive factor testing: an update. Appl Immunohistochem Mol Morphol. 2011 Dec;19(6):499-500. doi: 10.1097/PAI.0b013e31822a8eac. PMID 22089488
- [Background] Harbeck N, Sotlar K, Wuerstlein R, Doisneau-Sixou S. Molecular and protein markers for clinical decision making in breast cancer: today and tomorrow. Cancer Treat Rev. 2014 Apr;40(3):434-44. doi: 10.1016/j.ctrv.2013.09.014. Epub 2013 Sep 29. PMID 24138841
- [Background] Wazir U, Mokbel K. Emerging gene-based prognostic tools in early breast cancer: First steps to personalised medicine. World J Clin Oncol. 2014 Dec 10;5(5):795-9. doi: 10.5306/wjco.v5.i5.795. PMID 25493218
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Peto R, Davies C, Godwin J, Gray R, Pan HC, Clarke M, Cutter D, Darby S, McGale P, Taylor C, Wang YC, Bergh J, Di Leo A, Albain K, Swain S, Piccart M, Pritchard K. Comparisons between different polychemotherapy regimens for early breast cancer: meta-analyses of long-term outcome among 100,000 women in 123 randomised trials. Lancet. 2012 Feb 4;379(9814):432-44. doi: 10.1016/S0140-6736(11)61625-5. Epub 2011 Dec 5. PMID 22152853
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097
- [Background] Senkus E, Kyriakides S, Ohno S, Penault-Llorca F, Poortmans P, Rutgers E, Zackrisson S, Cardoso F; ESMO Guidelines Committee. Primary breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v8-30. doi: 10.1093/annonc/mdv298. No abstract available. PMID 26314782
- [Background] Gianni L, Dafni U, Gelber RD, Azambuja E, Muehlbauer S, Goldhirsch A, Untch M, Smith I, Baselga J, Jackisch C, Cameron D, Mano M, Pedrini JL, Veronesi A, Mendiola C, Pluzanska A, Semiglazov V, Vrdoljak E, Eckart MJ, Shen Z, Skiadopoulos G, Procter M, Pritchard KI, Piccart-Gebhart MJ, Bell R; Herceptin Adjuvant (HERA) Trial Study Team. Treatment with trastuzumab for 1 year after adjuvant chemotherapy in patients with HER2-positive early breast cancer: a 4-year follow-up of a randomised controlled trial. Lancet Oncol. 2011 Mar;12(3):236-44. doi: 10.1016/S1470-2045(11)70033-X. Epub 2011 Feb 25. PMID 21354370
- [Background] Slamon D, Eiermann W, Robert N, Pienkowski T, Martin M, Press M, Mackey J, Glaspy J, Chan A, Pawlicki M, Pinter T, Valero V, Liu MC, Sauter G, von Minckwitz G, Visco F, Bee V, Buyse M, Bendahmane B, Tabah-Fisch I, Lindsay MA, Riva A, Crown J; Breast Cancer International Research Group. Adjuvant trastuzumab in HER2-positive breast cancer. N Engl J Med. 2011 Oct 6;365(14):1273-83. doi: 10.1056/NEJMoa0910383. PMID 21991949
- [Background] Goldhirsch A, Gelber RD, Piccart-Gebhart MJ, de Azambuja E, Procter M, Suter TM, Jackisch C, Cameron D, Weber HA, Heinzmann D, Dal Lago L, McFadden E, Dowsett M, Untch M, Gianni L, Bell R, Kohne CH, Vindevoghel A, Andersson M, Brunt AM, Otero-Reyes D, Song S, Smith I, Leyland-Jones B, Baselga J; Herceptin Adjuvant (HERA) Trial Study Team. 2 years versus 1 year of adjuvant trastuzumab for HER2-positive breast cancer (HERA): an open-label, randomised controlled trial. Lancet. 2013 Sep 21;382(9897):1021-8. doi: 10.1016/S0140-6736(13)61094-6. Epub 2013 Jul 18. PMID 23871490
- [Background] Pivot X, Romieu G, Debled M, Pierga JY, Kerbrat P, Bachelot T, Lortholary A, Espie M, Fumoleau P, Serin D, Jacquin JP, Jouannaud C, Rios M, Abadie-Lacourtoisie S, Tubiana-Mathieu N, Cany L, Catala S, Khayat D, Pauporte I, Kramar A; PHARE trial investigators. 6 months versus 12 months of adjuvant trastuzumab for patients with HER2-positive early breast cancer (PHARE): a randomised phase 3 trial. Lancet Oncol. 2013 Jul;14(8):741-8. doi: 10.1016/S1470-2045(13)70225-0. Epub 2013 Jun 11. PMID 23764181
- [Background] Rodary C, Leplege A, Hill C. [Evaluation of the quality of life in clinical research in cancerology]. Bull Cancer. 1998 Feb;85(2):140-8. French. PMID 9752331
- [Background] Osoba D. What has been learned from measuring health-related quality of life in clinical oncology. Eur J Cancer. 1999 Oct;35(11):1565-70. doi: 10.1016/s0959-8049(99)00192-6. PMID 10673963
- [Background] de Haes J, Curran D, Young T, Bottomley A, Flechtner H, Aaronson N, Blazeby J, Bjordal K, Brandberg Y, Greimel E, Maher J, Sprangers M, Cull A. Quality of life evaluation in oncological clinical trials - the EORTC model. The EORTC Quality of Life Study Group. Eur J Cancer. 2000 May;36(7):821-5. doi: 10.1016/s0959-8049(00)00007-1. PMID 10785585
- [Background] Moinpour CM. Do quality of life assessments make a difference in the evaluation of cancer treatments? Control Clin Trials. 1997 Aug;18(4):311-7. doi: 10.1016/s0197-2456(97)00054-8. PMID 9257070
- [Background] Trask PC, Hsu MA, McQuellon R. Other paradigms: health-related quality of life as a measure in cancer treatment: its importance and relevance. Cancer J. 2009 Sep-Oct;15(5):435-40. doi: 10.1097/PPO.0b013e3181b9c5b9. PMID 19826365
- [Background] Johnson JR, Temple R. Food and Drug Administration requirements for approval of new anticancer drugs. Cancer Treat Rep. 1985 Oct;69(10):1155-9. PMID 4042094
- [Background] Gotay CC, Kawamoto CT, Bottomley A, Efficace F. The prognostic significance of patient-reported outcomes in cancer clinical trials. J Clin Oncol. 2008 Mar 10;26(8):1355-63. doi: 10.1200/JCO.2007.13.3439. Epub 2008 Jan 28. PMID 18227528
- [Background] Osoba D. Translating the science of patient-reported outcomes assessment into clinical practice. J Natl Cancer Inst Monogr. 2007;(37):5-11. doi: 10.1093/jncimonographs/lgm002. PMID 17951224
- [Background] Montazeri A. Quality of life data as prognostic indicators of survival in cancer patients: an overview of the literature from 1982 to 2008. Health Qual Life Outcomes. 2009 Dec 23;7:102. doi: 10.1186/1477-7525-7-102. PMID 20030832
- [Background] Quinten C, Coens C, Mauer M, Comte S, Sprangers MA, Cleeland C, Osoba D, Bjordal K, Bottomley A; EORTC Clinical Groups. Baseline quality of life as a prognostic indicator of survival: a meta-analysis of individual patient data from EORTC clinical trials. Lancet Oncol. 2009 Sep;10(9):865-71. doi: 10.1016/S1470-2045(09)70200-1. Epub 2009 Aug 18. PMID 19695956
- [Background] Braun DP, Gupta D, Grutsch JF, Staren ED. Can changes in health related quality of life scores predict survival in stages III and IV colorectal cancer? Health Qual Life Outcomes. 2011 Aug 3;9:62. doi: 10.1186/1477-7525-9-62. PMID 21812962
- [Background] Earlam S, Glover C, Fordy C, Burke D, Allen-Mersh TG. Relation between tumor size, quality of life, and survival in patients with colorectal liver metastases. J Clin Oncol. 1996 Jan;14(1):171-5. doi: 10.1200/JCO.1996.14.1.171. PMID 8558193
- [Background] Lis CG, Gupta D, Granick J, Grutsch JF. Can patient satisfaction with quality of life predict survival in advanced colorectal cancer? Support Care Cancer. 2006 Nov;14(11):1104-10. doi: 10.1007/s00520-006-0100-3. Epub 2006 Jul 4. PMID 16819630
- [Background] McKernan M, McMillan DC, Anderson JR, Angerson WJ, Stuart RC. The relationship between quality of life (EORTC QLQ-C30) and survival in patients with gastro-oesophageal cancer. Br J Cancer. 2008 Mar 11;98(5):888-93. doi: 10.1038/sj.bjc.6604248. Epub 2008 Feb 12. PMID 18268490
- [Background] Efficace F, Bottomley A, Coens C, Van Steen K, Conroy T, Schoffski P, Schmoll H, Van Cutsem E, Kohne CH. Does a patient's self-reported health-related quality of life predict survival beyond key biomedical data in advanced colorectal cancer? Eur J Cancer. 2006 Jan;42(1):42-9. doi: 10.1016/j.ejca.2005.07.025. Epub 2005 Nov 18. PMID 16298522
- [Background] Grande GE, Farquhar MC, Barclay SI, Todd CJ. Quality of life measures (EORTC QLQ-C30 and SF-36) as predictors of survival in palliative colorectal and lung cancer patients. Palliat Support Care. 2009 Sep;7(3):289-97. doi: 10.1017/S1478951509990216. PMID 19788770
- [Background] Maisey NR, Norman A, Watson M, Allen MJ, Hill ME, Cunningham D. Baseline quality of life predicts survival in patients with advanced colorectal cancer. Eur J Cancer. 2002 Jul;38(10):1351-7. doi: 10.1016/s0959-8049(02)00098-9. PMID 12091066
- [Background] Montgomery GH, Schnur JB, Kravits K. Hypnosis for cancer care: over 200 years young. CA Cancer J Clin. 2013 Jan;63(1):31-44. doi: 10.3322/caac.21165. Epub 2012 Nov 20. PMID 23168491
- [Background] Lang EV, Berbaum KS, Faintuch S, Hatsiopoulou O, Halsey N, Li X, Berbaum ML, Laser E, Baum J. Adjunctive self-hypnotic relaxation for outpatient medical procedures: a prospective randomized trial with women undergoing large core breast biopsy. Pain. 2006 Dec 15;126(1-3):155-64. doi: 10.1016/j.pain.2006.06.035. Epub 2006 Sep 7. PMID 16959427
- [Background] Montgomery GH, Weltz CR, Seltz M, Bovbjerg DH. Brief presurgery hypnosis reduces distress and pain in excisional breast biopsy patients. Int J Clin Exp Hypn. 2002 Jan;50(1):17-32. doi: 10.1080/00207140208410088. PMID 11778705
- [Background] Schnur JB, Bovbjerg DH, David D, Tatrow K, Goldfarb AB, Silverstein JH, Weltz CR, Montgomery GH. Hypnosis decreases presurgical distress in excisional breast biopsy patients. Anesth Analg. 2008 Feb;106(2):440-4, table of contents. doi: 10.1213/ane.0b013e31815edb13. PMID 18227298
- [Background] Liossi C, White P, Hatira P. A randomized clinical trial of a brief hypnosis intervention to control venepuncture-related pain of paediatric cancer patients. Pain. 2009 Apr;142(3):255-263. doi: 10.1016/j.pain.2009.01.017. Epub 2009 Feb 23. PMID 19231082
- [Background] Montgomery GH, Bovbjerg DH, Schnur JB, David D, Goldfarb A, Weltz CR, Schechter C, Graff-Zivin J, Tatrow K, Price DD, Silverstein JH. A randomized clinical trial of a brief hypnosis intervention to control side effects in breast surgery patients. J Natl Cancer Inst. 2007 Sep 5;99(17):1304-12. doi: 10.1093/jnci/djm106. Epub 2007 Aug 28. PMID 17728216
- [Background] Kamen C, Tejani MA, Chandwani K, Janelsins M, Peoples AR, Roscoe JA, Morrow GR. Anticipatory nausea and vomiting due to chemotherapy. Eur J Pharmacol. 2014 Jan 5;722:172-9. doi: 10.1016/j.ejphar.2013.09.071. Epub 2013 Oct 21. PMID 24157982
- [Background] Redd WH, Montgomery GH, DuHamel KN. Behavioral intervention for cancer treatment side effects. J Natl Cancer Inst. 2001 Jun 6;93(11):810-23. doi: 10.1093/jnci/93.11.810. PMID 11390531
- [Background] Montgomery GH, David D, Kangas M, Green S, Sucala M, Bovbjerg DH, Hallquist MN, Schnur JB. Randomized controlled trial of a cognitive-behavioral therapy plus hypnosis intervention to control fatigue in patients undergoing radiotherapy for breast cancer. J Clin Oncol. 2014 Feb 20;32(6):557-63. doi: 10.1200/JCO.2013.49.3437. Epub 2014 Jan 13. PMID 24419112
- [Background] Montgomery GH, Kangas M, David D, Hallquist MN, Green S, Bovbjerg DH, Schnur JB. Fatigue during breast cancer radiotherapy: an initial randomized study of cognitive-behavioral therapy plus hypnosis. Health Psychol. 2009 May;28(3):317-22. doi: 10.1037/a0013582. PMID 19450037
- [Background] Gregoire C, Bragard I, Jerusalem G, Etienne AM, Coucke P, Dupuis G, Lanctot D, Faymonville ME. Group interventions to reduce emotional distress and fatigue in breast cancer patients: a 9-month follow-up pragmatic trial. Br J Cancer. 2017 Nov 7;117(10):1442-1449. doi: 10.1038/bjc.2017.326. Epub 2017 Sep 19. PMID 28926526
- [Background] Bedard G, Zeng L, Zhang L, Lauzon N, Holden L, Tsao M, Danjoux C, Barnes E, Sahgal A, Poon M, Chow E. Minimal important differences in the EORTC QLQ-C30 in patients with advanced cancer. Asia Pac J Clin Oncol. 2014 Jun;10(2):109-17. doi: 10.1111/ajco.12070. Epub 2013 Apr 1. PMID 23551530
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735
- [Background] Zelen M. Randomized consent designs for clinical trials: an update. Stat Med. 1990 Jun;9(6):645-56. doi: 10.1002/sim.4780090611. PMID 2218168
- See also: 13th citation (pdf) — https://www.google.fr/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&ved=0ahUKEwiGreTb88rYAhUK7BQKHU0qBK4QFgguMAA&url=http%3A%2F%2Fwww.e-cancer.fr%2Fcontent%2Fdownload%2F148692%2F1867381%2Ffile%2FLes-cancers-en-France-edition-2015.pdf&usg=AOvVaw3SvYxld9y_1XzWhSyIEHS4
- See also: 27th citation — https://tel.archives-ouvertes.fr/tel-01234995/
- See also: 46th citation (pdf) — https://www.inserm.fr/sites/default/files/2017-11/Inserm_RapportThematique_EvaluationEfficaciteHypnose_2015.pdf